CLINICAL TRIAL: NCT02229526
Title: Randomised Clinical Trials of Fish Oil Supplementation in High Risk Pregnancies
Brief Title: Fish Oil Trials in Pregnancy for the Prevention of Pregnancy Complications ('FOTIP')
Acronym: FOTIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sjurdur Frodi Olsen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Sjurdur Frodi Olsen, Chief Physician, Centre-Leader, Centre for Fetal Programming, Denmark
Organization: Centre for Fetal Programming, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: DT2006-41-6257
Record Dates: First submitted 2014-03-03; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Preterm Birth; Intrauterine Growth Retardation; Pregnancy Induced Hypertension
Keywords: Fish oil supplementation; RCT; High risk pregnancies; Twin pregnancy; Preterm birth; Intrauterine growth retardation; Pregnancy induced hypertension
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation; Hypertension, Pregnancy-Induced | interventions — Fish Oils; Pikasol; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose fish oil (Active Comparator)
  Interventions: Dietary Supplement: Low dose fish oil
- Low dose olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: Low dose olive oil
- High dose fish oil (Experimental)
  Interventions: Dietary Supplement: High dose fish oil
- High dose olive oil (Placebo Comparator)
  Interventions: Dietary Supplement: High dose olive oil

INTERVENTIONS:
Dietary Supplement: Low dose fish oil — Four 1g gelatine capsules with fish oil (Pikasol: 32 % eicosapentaenoic acid (20:5n-3), 23 % docosahexaenoic acid (22:6n-3) and 2 mg tocopherol/ml)) corresponding to 2.7 g n-3 fatty acids per day.
  Other Names: Pikasol
  Arms: Low dose fish oil
Dietary Supplement: Low dose olive oil — Four 1 g capsules with olive oil (72 % oleic acid (18:1n-9) and 12 % linoleic acid (18:2n-6)) per day.
  Arms: Low dose olive oil
Dietary Supplement: High dose fish oil — Nine 1g gelatine capsules with fish oil (Pikasol: 32 % eicosapentaenoic acid (20:5n-3), 23 % docosahexaenoic acid (22:6n-3) and 2 mg tocopherol/ml)) corresponding to 6.1 g n-3 fatty acids per day.
  Other Names: Pikasol
  Arms: High dose fish oil
Dietary Supplement: High dose olive oil — Nine 1g gelatine capsules with olive oil (72 % oleic acid (18:1n-9) and 12 % linoleic acid (18:2n-6)) per day.
  Arms: High dose olive oil

SUMMARY:
The initial trial examined if fish oil supplementation during pregnancy could reduce the risk of pregnancy induced hypertension, intrauterine growth retardation, and preterm birth in pregnancies that were at increased risk of these complications. The study was designed as a multi-centre clinical trial based in 19 hospitals in seven countries in Europe.

ELIGIBILITY:
Inclusion Criteria:

* There were six subgroups with different inclusion criteria:
* The low dose (prophylactic) section enrolled women who after 16 weeks of gestation had been identified with an uncomplicated pregnancy, who in an earlier pregnancy had experienced preterm delivery (this was subgroup 1)
* Intrauterine growth retardation (subgroup 2) or pregnancy induced hypertension (subgroup 3)
* Women who had been identified with twin pregnancies (subgroup 4)
* The high dose ('therapeutic') section enrolled women with threatening pre-eclampsia (subgroup 5) or suspected intrauterine growth retardation in the current pregnancy (subgroup 6).

Exclusion Criteria:

* Diabetes mellitus in or before pregnancy
* Diagnosed severe fetal malformation or hydrops in current pregnancy
* Suspicion in current pregnancy, or occurrence in an earlier pregnancy, of placental abruption
* Drug or alcohol abuse
* Regular intake of fish oil or of non-steroidal antiinflammatory agents or other drugs with an effect on thombocyte function or eicosanoid metabolism
* Allergy to fish products.

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 1619 (Actual)
Dates: Start 1990-01; Primary Completion 1996-01 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy Induced Hypertension | Participants will be followed for the duration of pregnancy and the first few days after delivery, on average 20-26 weeks from recruitment and randomization.
  One or more recorded measurements of a diastolic blood pressure of above 90 mmHg at rest
Intrauterine growth retardation | Participants will be followed for the duration of pregnancy and the first few days after delivery, on average 20-26 weeks from recruitment and randomization.
  Birth weight below the 10th centile, as assessed from the infant's birth weight, gestational age and gender, on the basis of Danish standards (Br J Obstet Gynaecol 1986; 93: 128-134; and Acta Obstet Gynecol Scand 1985; 64: 65-70).
Preterm delivery | Participants will be followed for the duration of pregnancy and the first few days after delivery, on average 20-26 weeks from recruitment and randomization.
  Delivery at an estimated gestational age of less than 259 days (37 completed weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Niels J Secher, Professor, Principal Investigator — Rigshospitalet, Denmark; Sjurdur F Olsen, Professor, Principal Investigator — Center for Fetal Programming, Denmark

REFERENCES:
- [Result] Olsen SF, Secher NJ, Tabor A, Weber T, Walker JJ, Gluud C. Randomised clinical trials of fish oil supplementation in high risk pregnancies. Fish Oil Trials In Pregnancy (FOTIP) Team. BJOG. 2000 Mar;107(3):382-95. doi: 10.1111/j.1471-0528.2000.tb13235.x. PMID 10740336
- [Result] Olsen SF, Osterdal ML, Salvig JD, Weber T, Tabor A, Secher NJ. Duration of pregnancy in relation to fish oil supplementation and habitual fish intake: a randomised clinical trial with fish oil. Eur J Clin Nutr. 2007 Aug;61(8):976-85. doi: 10.1038/sj.ejcn.1602609. Epub 2007 Feb 7. PMID 17299499